CLINICAL TRIAL: NCT04907058
Title: Central Sleep Apnea Treated by CO2 Supplied by a Novel Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State Key Laboratory of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Yuan-Ming Luo, Proffessor, State Key Laboratory of Respiratory Disease
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202037
Record Dates: First submitted 2021-05-20; First posted 2021-05-28 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Central Sleep Apnea
Keywords: CSA
MeSH Terms: conditions — Sleep Apnea, Central

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with CO2 (Experimental): Patients were treated with an effective lowest concentration of CO2 delivered by the novel CO2 supply system.
  Interventions: Device: novel device with a comfortable mask

INTERVENTIONS:
Device: novel device with a comfortable mask — Using a device with a comfortable mask to supply constant low dose CO2 to treat patients.

SUMMARY:
In general, central sleep apnea is not as common as obstructive sleep apnea but it is common in patients with heart failure. It has been repeatedly shown that central sleep apnea worsens the prognosis of heart failure. The current concept in the development of CSA is hypocapnia which causes temporary cessation of respiratory neural output. Different methods for supplement of CO2 have been used to eliminate CSA. However, variation of CO2 concentration during overnight treatment and tight-fitting mask made the treatment uncomfortable. It is important to develop a device with a comfortable mask to supply constant low dose CO2 without breathing difficulty. We recently developed a device for treatment of CSA.

DETAILED DESCRIPTION:
Objective: To determine whether the device could improve sleep quality while eliminating CSA during the overnight study. Methods: Patients with central sleep apnea diagnosed by diaphragm EMG will be recruited in this study. CO2 concentration for treatment would be manually titrated during overnight PSG. Patients were then treated with an effective lowest concentration of CO2 derived from titration under PSG on the third night. The sleep apnea hypopnea index (AHI), central sleep apnea index (CHI), arousal index (ArI), Oxygen desaturation index (ODI), sleep structure, blood pressure, heart rate, diaphragm EMG, treatment side effects and treatment preference were to be observed.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to participate after informed consent
2. Males and females, any race and aged≥18yeras
3. Objectively confirmed central sleep apnea/Cheyne Stokes Respiration with an apnoea-hypopnoea- index (AHI)≥5/h by overnight polysomnography

Exclusion Criteria:

1. Obstructive sleep apnea
2. Severe COPD，FEV1/FVC<70% and FEV1<60%
3. Chronic CO2 retention with unknown reason
4. Severe nasal congestion
5. Poor understanding

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-23 (Actual)

PRIMARY OUTCOMES:
Apnea Hypopnea Index | One full night
  Total number of apneas and hypopneas/total sleep time (h)
Central sleep apnea index | One full night
  Total number of central sleep apneas/total sleep time (h)
Arousal Index | One full night
  Total number of arousals/total sleep time(h)
Oxygen Desaturation Index | One full night
  Total number of oxygen desaturations≥3% /total sleep time(h)
Sleep structure | One full night
  Assessment of the sleep efficiency (percentage is calculated by dividing Total Sleep Time by Total Time in bed)
Sleep structure | One full night
  Assessment of the sleep stage distribution (percentage calculated by diving the time of stage N1, N2, N3, NREM by total sleep time)
Adverse effects | One full night
  Using questionnaire named side effects of feeling to assess adverse effects exiting or not, including dyspnea, noise, bloating, itchy face, dry mouth, ophthalmalgia, stuffy nose, et al. When the side effect events in intervening condition 2 times more than baseline is worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanming Luo, PhD, Principal Investigator — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided